CLINICAL TRIAL: NCT07015125
Title: A Randomized Controlled Trial of a Transcutaneous Electrical Nerve Stimulation Device for the Acute Treatment of Migraine
Brief Title: Evaluation of a Wearable Device for Acute Treatment of Migraines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hinge Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1391996
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Migraine; Migraine With or Without Aura; Migraine, Acute; Migraine Headache
Keywords: Migraines; Acute Migraines; Headaches; Pain; Chronic Pain
MeSH Terms: conditions — Migraine Disorders; Headache; Pain; Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The study will be a randomized, controlled trial with a 3x3 factorial design (3 placements x 3 waveforms). Participants will be randomized to use the TENS device in one of three different placement locations. Each participant will test a total of 3 waveforms (two active waveforms and a sham waveform) in a randomized order over three distinct migraine episodes, with a 3-day washout period in between each treated migraine.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Center of Forehead (Experimental): Participants will use the TENS device on the center of the forehead. Participants use 2 active and 1 sham waveform in a randomized order to treat 3 distinct migraine episodes.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Side of Forehead (Experimental): Participants will use the TENS device on the side of the forehead. Participants use 2 active and 1 sham waveform in a randomized order to treat 3 distinct migraine episodes.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Back of Neck (Experimental): Participants will use the TENS device on the back of the neck. Participants use 2 active and 1 sham waveform in a randomized order to treat 3 distinct migraine episodes.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Use of TENS device for 1 hour during each migraine episode.
  Other Names: Enso

SUMMARY:
The goal of this clinical trial is to determine the efficacy of a new, improved neuromodulation device that can be worn on the head and neck to relieve migraine pain. To measure efficacy, investigators will compare how measured outcomes resulting from active stimulation with this device compare to those of sham treatment.

DETAILED DESCRIPTION:
The objective of this study is to examine the extent to which a transcutaneous electrical nerve stimulation (TENS) device safely helps participants with acute migraines reduce migraine pain intensity, achieve pain freedom, and experience sustained pain freedom. The TENS device attaches to a gel pad that can be worn in one of three placement locations to stimulate sensory nerves implicated in migraine pain. The TENS device outputs two active electrical waveforms that differ in stimulation intensity but can both be used to address migraine pain through a 1-hour treatment session. To achieve the study objective, investigators will perform a randomized controlled trial (RCT) with a 3x3 factorial design in which participants will be randomized across the 3 TENS device placement options and each participant will test 3 waveforms: two active waveforms and a sham waveform. Each waveform will be used in a distinct migraine episode. The investigators will evaluate the study aims for each active treatment (six in total) compared to its corresponding sham.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine with or without aura, identified via participant-provided medical records.
* Average migraine pain is 4 or more on the 0-10 Numerical Rating Scale (NRS) for pain.
* Passes ID-Migraine pre-screening questions and has ID-Migraine score ≥ 2:

  a. ID-Migraine pre-screening questions: i. How many headaches have participants experienced within the previous 3 months?
* Needs to be ≥ 6 headaches ii. Do the headaches that participants experience limit the ability to work, study, or enjoy life, or does the participant wish to speak with a healthcare professional about the headaches? (yes / no)
* Participant needs to respond "yes" b. ID-Migraine questions: i. Over the last 3 months, did participants have any of the following with headaches?
* Felt nauseated or sick to stomach (yes [1] / no [0])
* Light bothered them (a lot more than when headaches are not present)? (yes [1] / no [0])
* Headaches limited the ability to work, study, or do what needed to be done? (yes [1] / no [0])
* Able to understand and provide informed consent.
* Age 18 and older.
* US resident.
* Has experienced migraines for at least 1 year prior to recruitment.
* Onset of migraines occurred at age 50 years or younger.
* Average of at least 2 migraines per month of moderate to severe intensity.
* Is either on a) no medications or b) a stable dose of migraine-preventative medication for at least 2 months prior to recruitment.
* Willing to refrain from altering preventive medication for migraines (or from using botox), commit to using Enso as the first-line treatment, and wait at least 2 hours after Enso treatment before using any additional abortives during the study period.
* Participants must own an iPhone with iOS 15 or newer, or an Android phone with Android 9 or newer, with Bluetooth capability and access to either the Apple App Store (for iOS devices) or Google Play Store (for Android devices).
* Has an email account.

Exclusion Criteria:

* Typical migraine pain is < 4 out of 10 on the 0-10 NRS.
* Currently institutionalized.
* Currently is or has ever been a Hinge Health member.
* Use of antipsychotic medication up to 3 months before study recruitment.
* Diagnosis of cancer/malignant tumors in the last 5 years.
* Cognitive, behavioral, neurologic, or psychiatric disorder (e.g., dementia, Parkinson's, schizophrenia, stroke) that may interfere with the study or prevent the subject from complying with the requirements of the protocol.
* Has epilepsy.
* Has a history of major cardiovascular events such as strokes, arrhythmias, or myocardial infarction.
* Has a history of major migraine complications such as migrainous infarction or migraine aura-triggered seizure
* Diagnosed with secondary headache disorders including medication overuse headaches
* History of opioid, alcohol, or drug abuse in the last 1 year.
* Has a cardiac pacemaker, implanted defibrillator, spinal cord stimulator, pain pump, insulin pump, or any other implanted electronic device.
* Has a metal implant in the upper extremities or head.
* Has a history of major head or neck surgeries.
* Pregnant.
* Currently participating or has participated in a study with an investigational compound or device within the last 30 days before the screening visit.
* Currently using a TENS device to treat migraines.
* Received supraorbital nerve blocks or Botox treatment within 4 months prior to recruitment.
* Insufficient proficiency with the English language to take part in study procedures or complete online surveys.
* Planning to travel outside of the US within three months after consenting to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Safety/Adverse Events | Pre-treatment, 1, 2, and 24 hours post-treatment.
  Safety will be measured by comparing the number of reportable adverse events, with particular focus on serious adverse events, that occur for the 6 active treatments versus the corresponding sham. Adverse events will be assessed by asking participants of any symptoms or medical issues experienced since the last interaction or activity in the study. Participants will report details of the event, its circumstances, the severity, and outcome/resolution of the event in the post-treatment surveys. The events will be adjudicated by the Study Physician, who will determine seriousness, relatedness and reportability.
Pain Relief at 1 hour (Clinical Efficacy) | Pre-treatment, 1-hour post-treatment
  Pain relief will be measured by asking participants to report pain intensity using the 11-point Numeric Rating Scale (NRS) in the pre-treatment survey and in the post-treatment survey 1 hour after the initiation of treatment. NRS pain levels will be converted into categorical ratings of pain severity according to the following mapping between NRS and a 4-point Likert scale: (0-1 NRS => no pain; 2-3 NRS => mild pain; 4-6 NRS => moderate pain; 7-10 NRS => severe pain). Pain relief constitutes a change in pain level from severe or moderate pain to mild or no pain. The percentage of participants who achieve pain relief in the active and sham treatments will be compared. Six comparisons will be performed in total, for the 6 active treatments (3 placements x 2 active waveforms).

SECONDARY OUTCOMES:
Pain Relief at 2 hours | Pre-treatment, 2 hours post-treatment
  Pain relief will be measured by asking participants to report pain intensity using the 11-point Numeric Rating Scale (NRS) in the pre-treatment survey and in the post-treatment survey 2 hours after the initiation of treatment. NRS pain levels will be converted into categorical ratings of pain severity according to the following mapping between NRS and a 4-point Likert scale: (0-1 NRS => no pain; 2-3 NRS => mild pain; 4-6 NRS => moderate pain; 7-10 NRS => severe pain). Pain relief constitutes a change in pain level from severe or moderate pain to mild or no pain. The percentage of participants who achieve pain relief in the active and sham treatments will be compared. Six comparisons will be performed in total, for the 6 active treatments (3 placements x 2 active waveforms).
Pain Freedom at 2 hours | Pre-treatment, 1, 2 hours post-treatment.
  Pain freedom will be defined as a reduction in pain severity from mild, moderate, or severe at baseline to none at 2 hours, using the Numeric Rating Scale (NRS) mapped to a 4-point Likert scale, as based on literature. Six comparisons will be performed in total, for the 6 active treatments (3 placements x 2 active waveforms) vs the corresponding sham.
Sustained Pain Freedom | 24-hours post-treatment.
  Sustained pain freedom is defined as pain freedom at 24 hours without the use of anti-migraine medication or relapse during those 24 hours. Sustained pain freedom at 24 hours will be measured using the same four point Likert scale as used to measure pain freedom at 2 hours. Six comparisons will be performed in total, for the 6 active treatments (3 placements x 2 active waveforms) vs the corresponding sham.

CONTACTS AND LOCATIONS:
Overall Officials: Mallika Bariya, PhD, Principal Investigator — Hinge Health
Locations (1):
- Hinge Health, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No